CLINICAL TRIAL: NCT02237144
Title: Transfer Modality Research Initiative - Bangladesh
Acronym: TMRI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: International Food Policy Research Institute (Other)
Collaborators: United Nations World Food Programme (WFP) (Other); Federal Ministry of Economic Cooperation and Development (Germany) (Other Government); Swiss Agency for Development and Cooperation (Unknown); United States Agency for International Development (USAID) (U.S. Federal Agency); Department for International Development, United Kingdom (Other Government); Consortium of International Agricultural Research Centers (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Basic Science
Other Study IDs: AEARCTR-0000247
Record Dates: First submitted 2014-09-03; First posted 2014-09-11 (Estimated); Last update posted 2019-09-06 (Actual); Status verified 2019-09

CONDITIONS: Improving Pre-school Anthropometric Status; Improving Household Food Security; Improving Maternal Nutrition Knowledge
MeSH Terms: interventions — Food

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Cash transfer (Experimental): 1500 taka ($18.75) per household distributed monthly
  Interventions: Other: Cash transfer
- Food transfer (Experimental): 30 kg rice, 2 kg lentils, and 2 kg micro-nutrient fortified cooking oil per household distributed monthly
  Interventions: Other: Food transfer
- Food and cash transfer (Experimental): 15 kg of rice; 1 kg of lentils and 1 kg of micronutrient fortified cooking oil and 750 taka cash per household, distributed monthly
  Interventions: Other: Food and cash transfer
- Cash transfer + BCC (Experimental): 1500 taka ($18.75) per household distributed monthly Weekly, one hour meetings on maternal and child nutrition, sanitation and health knowledge, attitudes and practice Occasional home visits
  Interventions: Other: Cash transfer; Behavioral: Behavior Communication Change (BCC)
- Food transfer + BCC (Experimental): 30 kg rice, 2 kg lentils, and 2 kg micro-nutrient fortified cooking oil per household distributed monthly Weekly, one hour meetings on maternal and child nutrition, sanitation and health knowledge, attitudes and practice Occasional home visits
  Interventions: Other: Food transfer; Behavioral: Behavior Communication Change (BCC)

INTERVENTIONS:
Other: Cash transfer — 1500 taka ($18.75) per household distributed monthly
  Arms: Cash transfer; Cash transfer + BCC
Other: Food transfer — 30 kg rice, 2 kg lentils, and 2 kg micro-nutrient fortified cooking oil per household distributed monthly
  Arms: Food transfer; Food transfer + BCC
Other: Food and cash transfer — 15 kg of rice; 1 kg of lentils and 1 kg of micronutrient fortified cooking oil and 750 taka cash per household, distributed monthly
  Arms: Food and cash transfer
Behavioral: Behavior Communication Change (BCC) — Weekly, one hour meetings on maternal and child nutrition, sanitation and health knowledge, attitudes and practice Occasional home visits
  Arms: Cash transfer + BCC; Food transfer + BCC

SUMMARY:
This is a randomized control trial in two zones of Bangladesh (north and south). Treatment is assigned at the village level where treatments are: cash transfers (north and south); cash transfers + nutrition behavior communication change (north only); food transfers (north and south); food transfers + nutrition behavior communication change (south only); food-cash split (north and south); and controls (north and south). Within treatment localities, women living in very poor households are targeted to receive benefits for two years.

ELIGIBILITY:
Inclusion Criteria:

* Child age < 60 months

Exclusion Criteria:

* None

Ages: 15 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 5000 (Actual)
Dates: Start 2012-04; Primary Completion 2015-01 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Child anthropometry | Baseline. Up to 12 months. Up to 24 months.
  Height for age z scores Weight for height z scores Weight for age z scores Stunting Wasting Outcomes specified in terms of levels one year after intervention started (2013), two years after intervention started and as changes: 2012-2013, 2013-2014 and 2012-2014
Child food intake | Baseline. Up to 12 months. Up to 24 months.
  Number of unique foods consumed in previous 24 hours Number of food groups consumed in previous 24 hours Consumption of specified food groups - animal source foods, dairy, Vitamin A rich foods etc Caloric consumption in previous 24 hours Outcomes specified in terms of levels one year after intervention started (2013), two years after intervention started and as changes: 2012-2013, 2013-2014 and 2012-2014
Child health | Baseline. Up to 12 months. Up to 24 months.
  Did mother report child was ill in previous 2 weeks Outcomes specified in terms of levels one year after intervention started (2013), two years after intervention started and as changes: 2012-2013, 2013-2014 and 2012-2014
Distribution of food intake within the household | Baseline. Up to 12 months. Up to 24 months.
  Consumption of foods by all household members in previous 24 hours as recalled by mothers as measured by yes/no questions on foods, food groups and calories Outcomes specified in terms of levels one year after intervention started (2013), two years after intervention started and as changes: 2012-2013, 2013-2014 and 2012-2014
Household food security | Baseline. Up to 12 months. Up to 24 months.
  Food groups consumed by household in previous seven days Number of unique foods consumed in previous seven days Number of food groups consumed in previous seven days Number of food groups consumed in previous seven days weighted by nutritional value and frequency of consumption Value of food consumption in previous seven days Household caloric availability in previous seven days Outcomes specified in terms of levels one year after intervention started (2013), two years after intervention started and as changes: 2012-2013, 2013-2014 and 2012-2014
Maternal nutrition knowledge | Baseline. Up to 12 months. Up to 24 months.
  Maternal knowledge of infant and young child feeding practices (IYCF) Knowledge, attitudes, practice of IYCF Scored as yes/no and as a total score on all questions Levels assessed in 2013 and 2014 and as changes between 2012-2013, 2013-2014 and 2012-2014

SECONDARY OUTCOMES:
Household consumption | Baseline. Up to 12 months. Up to 24 months.
  Value of food consumption in previous seven days Value of monthly non-food consumption Value of monthly non-food consumption by specified sub-groups (clothing, medical expenses, education expenses, transport, consumables, semi-durables) Value of monthly household consumption (food and non-food) Outcomes specified in terms of levels one year after intervention started (2013), two years after intervention started and as changes: 2012-2013, 2013-2014 and 2012-2014
Household income | Baseline. Up to 12 months. Up to 24 months.
  Value of annual income derived from agriculture at endline (2014) Value of annual income derived from non-agricultural sources at endline (2014) Value of annual total income derived from all sources at endline (2014) Change in annual income (agriculture, non-agricultural, total) between 2012-2013, 2013-2014 and 2012-2014 Outcomes specified in terms of levels one year after intervention started (2013), two years after intervention started and as changes: 2012-2013, 2013-2014 and 2012-2014
Asset accumulation | Baseline. Up to 12 months. Up to 24 months.
  Index (z score) of consumer durables Index (z score) of productive assets Index of quality of housing stock Productive land ownership (ha) Outcomes specified in terms of levels one year after intervention started (2013), two years after intervention started and as changes: 2012-2013, 2013-2014 and 2012-2014
Women's empowerment | Up to 12 months. Up to 24 months.
  Index of women's decision making autonomy within the household Index of women's mobility outside the household Outcome measured as level in 2013, level in 2014 and change between 2013-2014
Information spillovers to non-beneficiaries | Up to 24 months.
  Knowledge of infant and young child feeding practices (IYCF) of mothers Knowledge, attitudes, practice of IYCF Scored as yes/no and as a total score on all questions Non-beneficiaries are mothers living near intervention households (within approximately a 10 minute walk) in the following treatment arms: North: cash, cash + BCC, control. South: food, food + BCC, control. Levels assessed in 2014

CONTACTS AND LOCATIONS:
Overall Officials: Akhter Ahmed, PhD, Principal Investigator — International Food Policy Research Institute; John Hoddinott, DPhil, Principal Investigator — International Food Policy Research Institute; Shalini Roy, PhD, Principal Investigator — International Food Policy Research Institute
Locations (1):
- International Food Policy Research Institute, Dhaka, Bangladesh

REFERENCES:
- [Derived] Hoddinott J, Ahmed I, Ahmed A, Roy S. Behavior change communication activities improve infant and young child nutrition knowledge and practice of neighboring non-participants in a cluster-randomized trial in rural Bangladesh. PLoS One. 2017 Jun 21;12(6):e0179866. doi: 10.1371/journal.pone.0179866. eCollection 2017. PMID 28636674